CLINICAL TRIAL: NCT06741917
Title: Comparison of the Post-operative Infection by Using Different Type Prophylactic Antibiotics in Low Risk Patients Who Underwent Retrograde Intrarenal Surgery
Brief Title: Retrograde Intrarenal Surgery Low Risk Trial
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 202405150MIND
Record Dates: First submitted 2024-12-08; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-07

CONDITIONS: Retrograde Intrarenal Surgery; Renal Stones
Keywords: retrograde intrarenal surgery; Prophylactic antibiotics
MeSH Terms: conditions — Nephrolithiasis | interventions — Levofloxacin; Cefmetazole; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oral Levofloxacin (Experimental)
  Interventions: Drug: Levofloxacin
- Intravenous cefmetzole (Active Comparator)
  Interventions: Drug: Cefmetazole (drug)

INTERVENTIONS:
Drug: Levofloxacin — single dose of oral Levofloxacin (500mg/tab) before retrograde intrarenal surgery
  Arms: Oral Levofloxacin
Drug: Cefmetazole (drug) — single dose of intravenous Cefmetazole (1000 mg)before retrograde intrarenal surgery
  Arms: Intravenous cefmetzole

SUMMARY:
In the treatment of kidney stones and upper ureteral stones, flexible ureteroscopic lithotripsy has become the mainstream choice due to its minimally invasive nature and high safety. However, there is still no universal consensus on the use of prophylactic antibiotics before surgery. Taiwan, located in the subtropical region, is one of the areas in the world with a high incidence of urinary tract stones. Currently, there are no established guidelines for the use of prophylactic antibiotics before flexible ureteroscopic lithotripsy in Taiwan. This study aims to evaluate the differences between single-dose, different types of prophylactic antibiotics in generally healthy adult patients undergoing flexible ureteroscopic lithotripsy.

DETAILED DESCRIPTION:
This study focuses on flexible ureteroscopic lithotripsy, a procedure commonly used to treat kidney stones and stones in the upper part of the ureter. This surgery is popular because it is minimally invasive and considered very safe. However, there is no clear agreement on whether or which antibiotics should be given to patients before the surgery to prevent infections.

Taiwan is one of the regions in the world with a high rate of urinary tract stones, and because of this, it is especially important to ensure that the best practices are followed to prevent infections during and after the surgery. Currently, there are no official guidelines in Taiwan on which antibiotics should be used before flexible ureteroscopic lithotripsy.

This study aims to compare different types of single-dose antibiotics given before the surgery to see if one is more effective than others in preventing infections. By looking at how different antibiotics perform, the study hopes to provide clearer guidance for doctors in choosing the best antibiotic treatment for patients, ultimately improving patient care and reducing the risk of infections after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Stone diameter < 3 cm or stone area < 900 mm2
* Preoperative(2 weeks) negative urine culture
* No active symptoms , including fever, dysuria, urinary frequency, urgency)
* Urinalysis WBC < 10/HPF

Exclusion Criteria:

* Immunocompromised
* Poor control Diabetes mellitus
* Allergy to antibiotics
* Ureteric stents or Foley catheter present
* Ureteric stricture
* Renal or urethral deformity
* Antibiotic treatment for urinary tract infection in the preceding 4 weeks

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Post-operative sepsis | Postoperative two weeks
  Postoperative systemic inflammatory response syndrome within two weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wollin DA, Joyce AD, Gupta M, Wong MYC, Laguna P, Gravas S, Gutierrez J, Cormio L, Wang K, Preminger GM. Antibiotic use and the prevention and management of infectious complications in stone disease. World J Urol. 2017 Sep;35(9):1369-1379. doi: 10.1007/s00345-017-2005-9. Epub 2017 Feb 3. PMID 28160088